CLINICAL TRIAL: NCT06275659
Title: An Exploratory Study to Evaluate a Digital Intervention to Disrupt Scratching in Atopic Dermatitis and Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Click Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CT-100-D-003
Record Dates: First submitted 2024-02-09; First posted 2024-02-23 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Psoriasis; Atopic Dermatitis
Keywords: Itching; DiNaMo
MeSH Terms: conditions — Psoriasis; Dermatitis, Atopic; Pruritus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- CT-100-004-A Psoriasis (Experimental)
  Interventions: Device: CT-100-004-A
- CT-100-004-B Psoriasis (Sham Comparator)
  Interventions: Device: CT-100-004-B
- CT-100-004-A Atopic Dermatitis (Experimental)
  Interventions: Device: CT-100-004-A
- CT-100-004-B Atopic Dermatitis (Sham Comparator)
  Interventions: Device: CT-100-004-B

INTERVENTIONS:
Device: CT-100-004-A — Digital Neuro-activation and Modulation (DiNaMo) component uses implicit training to strengthen inhibitory control. This intervention could help improve cognitive capabilities to help participants overcome the urge to scratch in response to an itch.
  Arms: CT-100-004-A Atopic Dermatitis; CT-100-004-A Psoriasis
Device: CT-100-004-B — The CT-100-D-004-B Processing speed training component uses implicit training targeting processing speed. This intervention could help improve cognitive capabilities to help participants overcome the urge to scratch in response to an itch.
  Arms: CT-100-004-B Atopic Dermatitis; CT-100-004-B Psoriasis

SUMMARY:
CT-100 is a platform that provides interactive, software based therapeutic components that may be used as part of a treatment in future software-based prescription digital therapeutics. One class of CT-100 components are Digital Neuro-activation and Modulation (DiNaMo TM) components.

DiNaMo components target key neural systems (including but not limited to systems related to sensory-, perceptual-, affective-, pain-, attention-, cognitive control, social- and self- processing) to optimally improve a participant's health.

DETAILED DESCRIPTION:
CT-100 is a platform that provides interactive, software based therapeutic components that may be used as part of a treatment in future software-based prescription digital therapeutics. One class of CT-100 components are Digital Neuro-activation and Modulation (DiNaMo TM) components.

DiNaMo components target key neural systems (including but not limited to systems related to sensory-, perceptual-, affective-, pain-, attention-, cognitive control, social- and self- processing) to optimally improve a participant's health.

The purpose of the proposed study is to evaluate initial effects of the DiNaMo component on measures of undesired behavior intensity and related outcomes in a variety of conditions, such as atopic dermatitis and psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Fluent in written and spoken English, confirmed by ability to read, understand and sign the informed consent form (ICF).
* Lives in the United States.
* Aged 18 years or older.
* Itch NRS ≥ 4 during screening.
* Meets indication-specific inclusion criteria (see Appendix 1), as reported by the study participant with adequate clinical documentation. (Documentation to be provided to the study team upon request.)
* Has an active email address and is willing and able to receive and respond to email messages.
* Has access to an internet connection during the study duration.
* Willing and able to comply with the study protocol and assessments.
* Is the sole user of an iPhone with an iPhone operating system (OS) 14 or later or a smartphone with an Android OS 10 or later for the duration of the study.
* Is willing and able to receive Short Message Service (SMS) text messages and notifications on their smartphone.

Exclusion Criteria:

* Pregnant or planning to become pregnant.
* Visual, dexterity or cognitive deficit so severe that it precludes the use of an App-based, reaction-time-based activity per investigator judgment.
* Severe psychiatric disorder involving a history of psychosis (e.g., schizophrenia, bipolar disorder or severe personality disorders).
* Psychiatric hospitalization in the past 6 months.
* Participation in any research study (including studies on psychotherapy, mindfulness, cognitive training or pharmacological treatment) during the past 3 months.
* Initiation or change in primary-disease-specific medication within 30 days prior to entering the study.
* Self-reported substance-use disorder within the past 1 year.
* Currently experiencing a skin infection.
* Planning the introduction of new therapies (including studies on psychotherapy, mindfulness, cognitive training or pharmacological treatment) during the 7-week study period.
* Anticipating a change in current pharmacological or psychotherapy treatment regimen during the 7-week study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Change in Peak Pruritus Numerical Rating Scale | Baseline to Week 4
  Change from baseline to Week 4 in the Peak Pruritus Numerical Rating Scale (PP-NRS)
Change in Dermatology Life Quality Index | Baseline to Week 4
  Change from baseline to Week 4 in the Dermatology Life Quality Index (DLQI)
Change in Quality of Life symptoms | Baseline to Week 4
  Change in QoL symptoms assessed with the PROMIS®-29+2 Profile v2.1 (PROMIS-29+2 Preference [PROPr]) scales (including mood, fatigue, pain interference, sleep, ability to participate in social functioning and cognitive function) from baseline to Week 4
Time in App | Baseline to Week 4
  Engagement with the App as measured by daily time in the App
Experience with Study App | Week 5
  Experience with the Study App as assessed by the User Experience Questionnaire after the Study App treatment period
Improved global rating of change | Baseline to Week 4
  Proportion of participants with an improvement as measured by the Global Rating of Change (GRC) score at Week 4

SECONDARY OUTCOMES:
Frequency of Adverse Events | Baseline to Week 5
  Frequency of adverse events (AEs)
Severity of Adverse Events | Baseline to Week 5
  Severity of adverse events (AEs)
Frequency of Serious Adverse Events | Baseline to Week 5
  Frequency of Serious Adverse Events (AEs)
Severity of Serious Adverse Events | Baseline to Week 5
  Severity of Serious Adverse Events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Shaheen Lakhan, Study Director — Click Therapeutics
Locations (1):
- Click Therapeutics, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No